CLINICAL TRIAL: NCT01962363
Title: A Phase 2A Clinical Trial of EPI-743 (Vincerinone™) on Visual Function in Friedreich's Ataxia Patients With Point Mutations
Brief Title: EPI-743 in Friedreich's Ataxia Point Mutations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Edison Pharmaceuticals Inc (Industry); Friedreich's Ataxia Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPI-743 PM
Record Dates: First submitted 2013-10-10; First posted 2013-10-14 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Friedreich's Ataxia
Keywords: Friedreich's ataxia point mutation
MeSH Terms: conditions — Friedreich Ataxia | interventions — alpha-tocotrienol quinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EPI-743 (Experimental): EPI-743, oral, 400mg three times daily for 3 months
  Interventions: Drug: EPI-743

INTERVENTIONS:
Drug: EPI-743 — EPI-743 (alpha-tocotrienol quinone) is a small molecule therapeutic that was rationally designed to replete reduced glutathione through NQO1-catalyzed electron transfer from NADPH.
  Other Names: Vincerinone, alpha-tocotrienol quinone

SUMMARY:
The purpose of this study is to evaluate the effects of EPI-743 in patients with Friedreich's Ataxia point mutations

DETAILED DESCRIPTION:
The primary objective of this study is to investigate whether treatment with EPI-743 has a discernible impact on visual function-including visual acuity, visual fields and color vision as well as on any of a number of functional and subject/clinician-rated scales relevant in the treatment of Friedreich's ataxia, and to determine the safety of treatment with EPI-743.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of genetically confirmed Friedreich's ataxia point mutation.
2. Visual acuity at baseline more than 15 letters on high contrast EDTRS at four meters.
3. FARS score of 20 to 90.
4. Male or female between 18 and 65 years of age.
5. Agreement to use contraception if within reproductive years
6. Hormone replacement therapy, if used, must remain stable for the duration of the study.
7. Willingness and ability to comply with study procedures.
8. Willingness and ability to arrive at study site metropolitan area day prior to evaluations.
9. Abstention from use of dietary supplements and non-prescribed medications at least 30 days prior to initiation of treatment and for the duration of the study. This would specifically include idebenone, Coenzyme Q10 and vitamin E.
10. Abstention from foods or beverages or bars fortified with Coenzyme Q10, vitamin E, super fortified functional foods or beverages at least 30 days prior to initiation of treatment and for the duration of the study.
11. Abstention from use of other investigative or non-approved drugs within 30 days of enrollment and for the duration of the study.
12. Subject can swallow multiple size 0 capsules.
13. Subject has voluntarily signed an IRB approved informed consent form to participate in the study after all relevant aspects of the study have been explained and discussed with the subject.

Exclusion Criteria:

1. Allergy to EPI-743 or sesame oil or nuts.
2. Clinically significant bleeding condition or abnormal PT/PTT INR (INR > two; PTT > two-times normal).
3. Liver insufficiency with LFTs greater than three-times upper normal limit at screening.
4. Renal insufficiency with creatinine > 1.5 at screening.
5. Fat malabsorption syndromes.
6. Any other respiratory chain diseases of the mitochondria or inborn errors of metabolism.
7. Any other ophthalmologic conditions.
8. Clinically significant cardiomyopathy with ejection fraction < 40 percent at screening.
9. Clinically significant arrhythmia within past two years requiring treatment.
10. Surgery planned through the duration of the study, including follow-up.
11. Pregnancy or breastfeeding.
12. Anticoagulant therapy within 30 days of enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Visual function | 3 months
  Low contrast acuity
Safety parameters | 3 months
  Clinical and laboratory safety parameters

SECONDARY OUTCOMES:
Visual function | 3 months
  Visual fields as assessed by Humphrey 30-2 exam; High contrast visual acuity
Neurologic function | 3 months
  Friedreich's Ataxia Rating Scale
Physical function | 3 months
  25-foot walk (for subjects capable of completing the test on enrollment);
Health related quality of life | 3 months
  Patient report via rating scale
Activities of Daily Living | 3 months
  Patient report via rating scale
Cardiac indices | 3 months
  Echocardiogram
Upper extremity function | 3 months
  9 hole peg test
Disease biomarkers | 3 months
  Glutathione cycle components

CONTACTS AND LOCATIONS:
Overall Officials: Theresa A Zesiewicz, MD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States